CLINICAL TRIAL: NCT02919982
Title: Benchmarking an Oral Anticoagulant Treatment Rate in Patients With Nonvalvular Atrial Fibrillation: A Study of Clinical Characteristics With Insight From Patient and Physician Perspectives
Brief Title: Benchmarking an Oral Anticoagulant Treatment Rate in Patients With Nonvalvular Atrial Fibrillation
Acronym: BOAT-AF
Status: Completed | Type: Observational
Sponsor: Baim Institute for Clinical Research (Other)
Collaborators: American College of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: AFP14
Record Dates: First submitted 2016-09-26; First posted 2016-09-30 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Nonvalvular Atrial Fibrillation
Keywords: Anticoagulant; Nonvalvular atrial fibrillation; Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish a benchmark for rate of prescription of oral anticoagulants (OA) in patients with non-valvular atrial fibrillation (NVAF) seen in an ambulatory care setting, based on independent medical assessment of clinical data and physician and patient surveys. The study will also assess reasons for not prescribing OA to prevent thromboembolic complications in patients with NVAF seen in ambulatory care, and patients' perspectives of non-use of OA for treatment of NVAF.

DETAILED DESCRIPTION:
At participating centers within the American College of Cardiology's (ACC) PINNACLE Registry, patients with nonvalvular atrial fibrillation who, according to ACC guidelines, are indicated as having an indication for oral anticoagulants (OA), but who are not receiving them, will be identified. Recruitment of participating physicians will also take place through collaboration with the PINNACLE Registry. Physician and patient participants will be asked to complete clinical surveys characterizing use and perception of OA therapy for each individual patient. The Baim Institute for Clinical Research (Baim Institute) serves as an analytic center for the PINNACLE Registry and will collaboratively lead this project with the ACC. The information collected from the PINNACLE Registry will include patient characteristics, site characteristics (volume, region, etc.) and the treating physician characteristics. Information from the patient and physician surveys will provide the clinical reasons for prior nontreatment as assessed by the treating physicians as well as the patients' perception of OA treatment (overall and according to pre-specified subgroups based on patient and site characteristics). Information will also be gathered from the patients' chart.

The above data will be compiled and reviewed by a committee of cardiologists who will assess whether OA treatment would be appropriate based on all the clinical factors assessed.

The BOAT-AF data will be linked to data from the PINNACLE Registry for the patients for whom surveys have been collected. Linking the two datasets will allow assessment of whether or not the participating physicians prescribed OA treatment and whether those patients started OA treatment within approximately 12 months after completing the questionnaire.

ELIGIBILITY:
Inclusion Criteria: A patient must meet all of the following criteria to participate in this study:

* Able and willing to complete the survey;
* Diagnosed with nonvalvular atrial fibrillation and CHA2DS2-VASc ≥ 2;
* Not currently treated with oral anticoagulants according to the PINNACLE Registry data;
* Enrolled in the PINNACLE Registry;
* Last physician office visit within the prior 18 months; and
* Age ≥ 18 years.

Exclusion Criteria: A patient will be excluded from participating in the study for any of the following reasons:

* Patient is no longer being followed at the local practice;
* Patient declines participation; and/or
* Patient is unable to speak or read English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes, from participating centers within the PINNACLE Registry, patients with nonvalvular atrial fibrillation identified as having an indication for oral anticoagulants, according to guidelines developed by the American College of Cardiology, but not receiving them.
Sampling Method: Non-Probability Sample
Enrollment: 817 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
A benchmark rate of OA treatment in patients with NVAF | Baseline
  This rate of OA will be based on assessment of appropriateness of OA treatment based on clinical guidelines by cardiologists using clinical data and the physician and patient surveys.

SECONDARY OUTCOMES:
Physician Reason for not prescribing OA; Patient perspectives on non-use of OA | Baseline
  Information from the patient and physician surveys will provide the clinical reasons for prior nontreatment as assessed by the treating physicians as well as the patients' perception of OA treatment (overall and according to pre-specified subgroups based on patient and site characteristics). Information will also be gathered from the patients' charts.

OTHER OUTCOMES:
Change in rate of OA use | 1 year
  Via linking the BOAT-AF data with the PINNACLE Registry data, we will assess if there is a change in the rate of OA one year following the BOAT-AF surveys

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Cannon, MD, Principal Investigator — Baim Institute for Clinical Research
Locations (21):
- United States (21):
  - Alaska Heart Institute, Anchorage, Alaska
  - Orange County Heart Institute and Research Center, Orange, California
  - Clearwater Cardiovascular & Interventional Consultants MD PA, Clearwater, Florida
  - Holy Cross Hospital, Inc., Fort Lauderdale, Florida
  - Heartwell LLP, Miami, Florida
  - Cardiac Institute of the Palm Beaches, Palm Beach Gardens, Florida
  - Adventist Health Partners, Inc. Amita Health, Hinsdale, Illinois
  - Delmarva Heart LLC, Salisbury, Maryland
  - Michigan Heart - St. Joseph Mercy Health System, Ann Arbor, Michigan
  - Munson Medical Group, Traverse City, Michigan
  - CardioCare, PC, Hillsborough, New Jersey
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Southern Oregon Cardiology, Medford, Oregon
  - Cardiology Consultants of Philadelphia - Lansdale, Lansdale, Pennsylvania
  - The Heart Institute of East Texas, Lufkin, Texas
  - Waco Cardiology Associates, Waco, Texas
  - Revere Health-Heart of Dixie Cardiology Central Utah Clinic PC, St. George, Utah
  - Centra Health, Inc. dba Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Western Washington Medical Group, Inc., Everett, Washington
  - Kootenai Health dba Heart Clinics of the Northwest, Spokane, Washington